CLINICAL TRIAL: NCT01094912
Title: Procedures of Locoregional Analgesia and Quality of Life in Palliative Care
Brief Title: Procedures of Locoregional Analgesia and Quality of Life in Palliative Care Units
Acronym: TALViSoP
Status: Suspended | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Limoges (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: I08014/TALViSoP
Record Dates: First submitted 2010-03-26; First posted 2010-03-29 (Estimated); Last update posted 2015-09-01 (Estimated); Status verified 2015-03

CONDITIONS: Pain
Keywords: Cancer pain
MeSH Terms: conditions — Pain; Cancer Pain | interventions — Analgesics, Opioid

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: opioids

SUMMARY:
Number of patients in mobile palliative care units have pain of both nociceptive and neuropathic origin. In certain cases, procedures of locoregional analgesia can be helpful.

The Purpose of this study is to evaluate the impact of techniques of locoregional analgesia in a palliative population

DETAILED DESCRIPTION:
Cancer pain is a serious problem in the palliative population. In particular, pain due to compression or invasion of nerve tissue by metastasis is frequent and often unresponsive to oral drug therapy and even to epidural administration of opioids. In such refractory pain in a palliative setting, one modality that could be helpful is the use of technics of locoregional analgesia. Currently, they are routinely used for the management of acute postoperative pain and become to be more widely used for cancer surgery. For example, intrapleural intercostal nerve blocks after major lung resection or preincisional paravertebral blocks after breast surgery have been shown to improve pain control. However, locoregional analgesia is only occasionally used in chronic cancer pain.

The procedures used are epidural analgesia, rachianesthesia, or continuous nerve blocks. L-bupivacaine will be used. The procedure will be performed only if the injection test is positive.

The patients will be evaluated before and after the procedure, the patient being his/her own control. Evaluations will take place immediately before the procedure, then at 48 hours, 1 week and 1 month after the procedure.

ELIGIBILITY:
Inclusion Criteria:

* Patient ≥ 18 years-old, male or female, whatever his/her ethnic group
* Patient with untreatable cancer
* Patient hospitalized in a palliative care unit, with a life expectancy ≥ 1 week
* Pain unresponsive to conventional treatments
* Effectiveness of the injection test
* Signed informed consent

Exclusion Criteria:

* Patients > 18 years-old
* Patients with pain other than cancer pain
* Patient's refusal
* Coagulation disorders
* Local infection
* Known hypersensitivity to local analgesics
* Inefficacy of the injection test.
* Contraindication for analgesics

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Estimated)
Dates: Start 2010-04; Primary Completion 2015-10 (Estimated); Study Completion 2015-10 (Estimated)

PRIMARY OUTCOMES:
Change in patients global quality of life | 1 week after first injection
  To evaluate the change in patients global quality of life, assessed by the item 15 of the validated quality of life scale EORTC QLQ-C15 PAL. Evaluations will take place before the procedure of locoregional analgesia and 1 week after.

SECONDARY OUTCOMES:
change in patient's global quality of life | 2 days and 1 week after procedure
  * evaluate the change in EORTC QLQ-C15 PAL score, assessed before the procedure of locoregional analgesia and 1 week after.
  * evaluate the change in patient's global quality of life, assessed by the item 15 of the validated quality of life scale EORTC QLQ-C15 PAL at 48 hours and 1 week post-procedure.
  * evaluate pain at 48 hours post-procedure
  * evaluate the change in doses of conventional treatments at 1 week

CONTACTS AND LOCATIONS:
Overall Officials: Gérard TERRIER, MD, Study Chair — CHU Limoges
Locations (6):
- France (6):
  - Centre Hospitalier Universitaire - Hôpital Saint André, Bordeaux
  - Centre Hospitalier de Châteauroux, Châteauroux
  - Centre Hospitalier de Guéret, Guéret
  - CHU Limoges, Liomges
  - Centre Hospitalier Local, Saint-Léonard-de-Noblat
  - Centre Hospitalier de Tulle, Tulle